CLINICAL TRIAL: NCT05566509
Title: Physical Activity and Balance Changes in Operated Patients Because of Breast Cancer
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Other Study IDs: SaglikBilimleriUEZBERCI
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Balance and Physical Activity Deficits After Breast Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast Conservative Surgery: The patients who had minimally invasive surgery.
  Interventions: Procedure: Breast excision
- Mastectomy: The patients who had invasive and destructive surgery.
  Interventions: Procedure: Breast excision

INTERVENTIONS:
Procedure: Breast excision — some patient had minimal excision, some had maximal excision.

SUMMARY:
Balance and physical activity deficits are theoretically expected in patients operated on for breast cancer. A significant decrease in the physical activity occurred, Their balance did not deteriorate in the follow-ups. This was independent of the type of the surgery performed.

ELIGIBILITY:
Inclusion Criteria:

* patients who had breast cancer surgery

Exclusion Criteria:

* balance disorders, physical disability that will affect balance (polio sequelae) and neurological diseases with balance system and/or peripheral nervous system involvement (diabetic neuropathy and familial/genetic neuropathies, Parkinson's Disease, Multiple Sclerosis, Alzheimer's Disease), bone metastasis, patients who have undergone reconstructive surgery

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — woman breast cancer
Study Population: breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
decrease in the physical activity | 2
  Balance and physical activity deficits are theoretically expected in patients operated on for breast cancer.

IPD SHARING:
Plan to Share IPD: Undecided